CLINICAL TRIAL: NCT00209638
Title: Phase I/II Study of Oral S-1 Plus Irinotecan in Patients With Advanced Gastric Cancer: Hokkaido Gastrointestinal Cancer Study Group HGCSG0101
Brief Title: Phase I/II Study of Oral S-1 Plus Irinotecan in Patients With Advanced Gastric Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hokkaido Gastrointestinal Cancer Study Group (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGCSG0002
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2006-04-21 (Estimated); Status verified 2006-04

CONDITIONS: Gastric Cancer
Keywords: Irinotecan,; S-1,; Phase I/II,; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan; S 1 (combination)

INTERVENTIONS:
Drug: irinotecan
Drug: S-1

SUMMARY:
To assess the usefulness of irinotecan plus S-1 therapy based on the antitumor effect and survival period. by performing a phase I/II study of this combination in patients with inoperable or with postoperative gastric cancer

DETAILED DESCRIPTION:
A multicenter Open-label, single-arm, phase I/II clinical trial is conducted on patients with histological stage IV gastric cancer given irinotecan plus S-1. The usefulness of this regimens as 1st line therapy for gastric cancer was evaluated by the disease-free survival rate (DFR), overall survival rate (OS), incidence and severity of adverse event.

ELIGIBILITY:
Inclusion Criteria:

・ Eligibility criteria

1. Histological diagnosis of gastric adenocarcinoma.
2. Measurable or assessable lesions.
3. Age: 18 ~ 75 years.
4. Performance Status (ECOG): 0 ~ 2.
5. No prior chemotherapy or only one regimen of previous chemotherapy (with a washout period >4 weeks after the final day of the previous therapy). Adjuvant chemotherapy is not defined as previous therapy.
6. No history of treatment with CPT-11 or S-1.
7. No history of radiotherapy to the abdomen.
8. Oral intake of S-1 is possible.
9. Adequate function of major organs (bone marrow, heart, lungs, liver etc.). WBC 3,500/mm3 and 12,000/mm3. Hb 10.0 g/dl. Platelet count 100,000/mm3. GOT and GPT 2.5times the upper limit of normal (excluding liver metastasis). T-Bil 2.0mg/dl. Creatinine <1.5 mg/dl (but if it is 1.0 ~ 1.5 mg/dl, the dose of S-1 can be decreased according to the dose reduction criteria to allow registration in the trial). Normal ECG (not considering clinically unimportant arrhythmias and ischemic changes).
10. Predicted survival for >3 months.
11. Able to give written informed consent

Exclusion Criteria:

1. Severe pleural effusion or ascites.
2. Metastasis to the central nervous system (CNS).
3. Active gastrointestinal bleeding.
4. Active infection.
5. Diarrhea (watery stools).
6. Uncontrolled ischemic heart disease.
7. Serious complications (such as intestinal paralysis, intestinal obstruction, interstitial pneumonia or pulmonary fibrosis, uncontrolled diabetes mellitus, heart failure, renal failure, or hepatic failure).
8. Active multiple cancer.
9. Severe mental disorder.
10. Pregnancy, possible pregnancy, or breast-feeding.
11. Flucytosine treatment
12. Gilbert's syndrome.
13. Judged to be ineligible for this protocol by the attending physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2000-05; Study Completion 2003-04

PRIMARY OUTCOMES:
objective tumor response

SECONDARY OUTCOMES:
Response duration, time to progression, overall survival, and safety will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Asaka, MD, PhD, Study Chair — Hokkaido Gastrointestinal Cancer Study Group